CLINICAL TRIAL: NCT00509795
Title: A Randomized, Double Masked, Active Controlled Phase III Study of the Efficacy, Safety, and Tolerability of Repeated Doses of Intravitreal VEGF Trap in Subjects With Neovascular Age-Related Macular Degeneration
Brief Title: Vascular Endothelial Growth Factor VEGF Trap-Eye:Investigation of Efficacy and Safety in Wet Age-Related Macular Degeneration(AMD)
Acronym: VIEW1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VGFT-OD-0605
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Results first posted 2012-04-16 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ranibizumab 0.5mg Q4 (Active Comparator)
  Interventions: Biological: ranibizumab
- aflibercept injection 2.0mg Q4 (Experimental)
  Interventions: Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321)
- aflibercept injection 0.5mg Q4 (Experimental)
  Interventions: Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321)
- aflibercept injection 2.0mg Q8 (Experimental)
  Interventions: Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Biological: ranibizumab — Participants received a 0.5mg dose of ranibizumab via intravitreal (IVT) injection every 4 weeks for the first year. Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
  Other Names: Lucentis
  Arms: ranibizumab 0.5mg Q4
Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321) — Participants received a 2.0mg dose of aflibercept injection every 4 weeks for the first year. Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
  Other Names: VEGF Trap-Eye; BAY86-5321
  Arms: aflibercept injection 2.0mg Q4
Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321) — Participants received a 0.5mg dose of aflibercept injection every 4 weeks for the first year. Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
  Other Names: VEGF Trap-Eye; BAY86-5321
  Arms: aflibercept injection 0.5mg Q4
Biological: aflibercept injection (VEGF Trap-Eye, BAY86-5321) — Participants received a 2.0mg dose of aflibercept injection every 8 weeks (including one additional 2.0 mg dose at Week 4) for the first year and were to receive sham injections at interim monthly visits. Thereafter a dose may be administered as frequently as every 4 weeks, but no less frequently than every 12 weeks.
  Other Names: VEGF Trap-Eye; BAY86-5321
  Arms: aflibercept injection 2.0mg Q8

SUMMARY:
This study is a phase 3, double-masked, randomized, study of the efficacy and safety of VEGF Trap-Eye in patients with neovascular age-related macular degeneration. Approximately 1200 patients will be randomized in the US and Canada.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent.
2. Men and women ≥ 50 years of age.
3. Active primary or recurrent subfoveal CNV lesions secondary to AMD, including juxtafoveal lesions that affect the fovea as evidenced by FA in the study eye.
4. Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) of: letter score of 73 to 25 (20/40 to 20/320) in the study eye at 4 meters.
5. Willing, committed, and able to return for ALL clinic visits and complete all study-related procedures.
6. Able to read, (or, if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent or a family member. See Appendix J.4) understand and willing to sign the informed consent form.

Key

Exclusion Criteria:

1. Any prior ocular (in the study eye) or systemic treatment or surgery for neovascular AMD except dietary supplements or vitamins.
2. Any prior or concomitant therapy with another investigational agent to treat neovascular AMD in the study eye, except dietary supplements or vitamins.
3. Any prior treatment with anti-VEGF agents in the study eye.
4. Total lesion size > 12 disc areas (30.5 mm^2, including blood, scars and neovascularization) as assessed by FA in the study eye.
5. Subretinal hemorrhage that is either 50% or more of the total lesion area, or if the blood is under the fovea and is 1 or more disc areas in size in the study eye. (If the blood is under the fovea, then the fovea must be surrounded 270 degrees by visible CNV.)
6. Scar or fibrosis, making up > 50% of total lesion in the study eye.
7. Scar, fibrosis, or atrophy involving the center of the fovea.
8. Presence of retinal pigment epithelial tears or rips involving the macula in the study eye.
9. History of any vitreous hemorrhage within 4 weeks prior to Visit 1 in the study eye.
10. Presence of other causes of CNV in the study eye.
11. History or clinical evidence of diabetic retinopathy, diabetic macular edema or any other vascular disease affecting the retina,other than AMD, in either eye.
12. Prior vitrectomy in the study eye.
13. History of retinal detachment or treatment or surgery for retinal detachment in the study eye.
14. Any history of macular hole of stage 2 and above in the study eye.
15. Any intraocular or periocular surgery within 3 months of Day 1 on the study eye, except lid surgery, which may not have taken place within 1 month of day 1, as long as its unlikely to interfere with the injection.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1217 (Actual)
Dates: Start 2007-08; Primary Completion 2010-09 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vitti, MD, Study Director — Regeneron Pharmaceuticals
Locations (157):
- United States (147):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Beverly Hills, California
  - Campbell, California
  - Fullerton, California
  - Glendale, California
  - Irvine, California
  - La Jolla, California
  - Loma Linda, California
  - Los Angeles, California
  - Menlo Park, California
  - Mountain View, California
  - Oakland, California
  - Palm Springs, California
  - Pasadena, California
  - Poway, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Santa Ana, California
  - Torrance, California
  - Ventura, California
  - Westlake Village, California
  - Yorba Linda, California
  - Aurora, Colorado
  - Denver, Colorado
  - Bridgeport, Connecticut
  - Hamden, Connecticut
  - New Haven, Connecticut
  - New London, Connecticut
  - Altamonte Springs, Florida
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Mt. Dora, Florida
  - Orlando, Florida
  - Oscala, Florida
  - Palm Beach Gardens, Florida
  - Pensacola, Florida
  - Sarasota, Florida
  - Stuart, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Honolulu, Hawaii
  - ‘Aiea, Hawaii
  - Oak Brook, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - New Albany, Indiana
  - Iowa City, Iowa
  - Wichita, Kansas
  - Louisville, Kentucky
  - Paducah, Kentucky
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Bangor, Maine
  - Portland, Maine
  - Baltimore, Maryland
  - Chevy Chase, Maryland
  - Hagerstown, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Peabody, Massachusetts
  - Ann Arbor, Michigan
  - Battle Creek, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Jackson, Michigan
  - Royal Oak, Michigan
  - Southfield, Michigan
  - West Bloomfield, Michigan
  - Edina, Minnesota
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Florissant, Missouri
  - Kansas City, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Lawrenceville, New Jersey
  - New Brunswick, New Jersey
  - Northfield, New Jersey
  - Teaneck, New Jersey
  - Toms River, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - Lynbrook, New York
  - New York, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - Slingerlands, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Southern Pines, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Ashland, Oregon
  - Portland, Oregon
  - Salem, Oregon
  - Kingston, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsberg, Pennsylvania
  - Pittsburgh, Pennsylvania
  - West Mifflin, Pennsylvania
  - Wyomissing, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greenville, South Carolina
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - Corpus Cristi, Texas
  - Dallas, Texas
  - DeSoto, Texas
  - Fort Worth, Texas
  - Galveston, Texas
  - Houston, Texas
  - McAllen, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Charlottesville, Virginia
  - Fairfax, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Silverdale, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Canada (10):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Halifax, Nova Scotia
  - London, Ontario
  - Mississauga, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Regina, Saskatchewan

REFERENCES:
- [Derived] Li E, Donati S, Lindsley KB, Krzystolik MG, Virgili G. Treatment regimens for administration of anti-vascular endothelial growth factor agents for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2020 May 5;5(5):CD012208. doi: 10.1002/14651858.CD012208.pub2. PMID 32374423
- [Derived] Moshfeghi DM, Thompson D, Saroj N. Changes in neovascular activity following fixed dosing with an anti-vascular endothelial growth factor agent over 52 weeks in the phase III VIEW 1 and VIEW 2 studies. Br J Ophthalmol. 2020 Sep;104(9):1223-1227. doi: 10.1136/bjophthalmol-2019-315021. Epub 2019 Dec 11. PMID 31826853
- [Derived] Yuzawa M, Fujita K, Wittrup-Jensen KU, Norenberg C, Zeitz O, Adachi K, Wang EC, Heier J, Kaiser P, Chong V, Korobelnik JF. Improvement in vision-related function with intravitreal aflibercept: data from phase 3 studies in wet age-related macular degeneration. Ophthalmology. 2015 Mar;122(3):571-8. doi: 10.1016/j.ophtha.2014.09.024. Epub 2014 Nov 6. PMID 25439429

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 164 sites in the United States and Canada. Recruitment period: 02 Aug 2007 to 15 Sep 2009.
Pre-assignment Details: 2063 patients were screened, 1217 randomized, and 1215 included in the Safety Analysis Set (SAF). The Full Analysis Set (FAS) included 1210 patients with at least 1 post-baseline assessment. The Per Protocol Set (PPS) included 1089 patients who received ≥ 9 doses of study drug and attended ≥ 9 scheduled visits during the first year.
Groups:
- Ranibizumab 0.5mg Q4: Patients received a 0.5mg dose of ranibizumab via intravitreal (IVT) injection every 4 weeks for the first year.
- IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4: Patients received a 2.0mg dose of Intravitreal Aflibercept Injection (IAI, EYLEA, VEGF Trap-Eye) every 4 weeks for the first year.
- IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4: Patients received a 0.5mg dose of Intravitreal Aflibercept Injection (IAI, EYLEA, VEGF Trap-Eye) every 4 weeks for the first year.
- IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8: Patients received a 2.0mg dose of Intravitreal Aflibercept Injection (IAI, EYLEA, VEGF Trap-Eye) every 8 weeks (including one additional 2.0 mg dose at Week 4) for the first year and received sham injections at interim monthly visits.
Period: Overall Study
Arm/Group | Ranibizumab 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8
Started | 306 | 304 | 304 | 303
Patients Received Treatment (SAF) | 304 | 304 | 304 | 303
Full Analysis Set (FAS) Population | 304 | 304 | 301 | 301
Per Protocol Set (PPS) Population | 269 | 285 | 270 | 265
Completed | 284 | 293 | 277 | 276
Not Completed | 22 | 11 | 27 | 27
Not completed — Adverse Event | 4 | 3 | 5 | 4
Not completed — Death | 3 | 1 | 2 | 7
Not completed — Lack of Efficacy | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 4 | 4
Not completed — OTHER | 1 | 0 | 4 | 1
Not completed — Protocol Violation | 3 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 10 | 5 | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Ranibizumab 0.5mg Q4: Patients received a 0.5mg dose of ranibizumab via IVT injection every 4 weeks for the first year.
- IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8: Patients received a 2.0mg dose of Intravitreal Aflibercept Injection (IAI, EYLEA, VEGF Trap-Eye) every 8 weeks (including one additional 2.0 mg dose at Week 4) for the first year and were to receive sham injections at interim monthly visits.
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8 | Total
Number analyzed (Participants) | 304 | 304 | 304 | 303 | 1215
Age Continuous [Mean (Standard Deviation); unit: years] — SAF population used for analysis.
  years | 78.2 (7.59) [0 to 0] | 77.7 (7.93) [0 to 0] | 78.3 (8.10) [0 to 0] | 77.9 (8.39) [0 to 0] | 78.0 (8.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 194 | 169 | 179 | 714
  Male | 132 | 110 | 135 | 124 | 501
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — SAF population used for analysis.
  Participants
    Hispanic or Latino | 7 (0) [0 to 0] | 11 (0) [0 to 0] | 11 (0) [0 to 0] | 12 (0) [0 to 0] | 41
    Not Hispanic or Latino | 297 | 293 | 293 | 291 | 1174
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — SAF population used for analysis.
  Participants
    American Indian or Alaska Native | 2 (0) [0 to 0] | 0 (0) [0 to 0] | 2 (0) [0 to 0] | 1 (0) [0 to 0] | 5
    Asian | 0 (0) [0 to 0] | 3 (0) [0 to 0] | 5 (0) [0 to 0] | 4 (0) [0 to 0] | 12
    Native Hawaiian or Other Pacific Islander | 1 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 1 (0) [0 to 0] | 2
    Black or African American | 1 (0) [0 to 0] | 1 (0) [0 to 0] | 0 (0) [0 to 0] | 1 (0) [0 to 0] | 3
    White | 296 (0) [0 to 0] | 295 (0) [0 to 0] | 294 (0) [0 to 0] | 289 (0) [0 to 0] | 1174
    More than one race | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 0 (0) [0 to 0] | 1 (0) [0 to 0] | 1
    Unknown or Not Reported | 4 (0) [0 to 0] | 5 (0) [0 to 0] | 3 (0) [0 to 0] | 6 (0) [0 to 0] | 18
Baseline National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) total score [Mean (Standard Deviation); unit: scores on a scale] — SAF population used for analysis. The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales which are all scored from 0-100. To reach the overall composite score, each sub-scale score is averaged in order to give each sub-scale equal weight.
  scores on a scale | 71.7 (17.29) [0 to 0] | 70.4 (16.60) [0 to 0] | 71.1 (17.72) [0 to 0] | 69.5 (16.82) [0 to 0] | 70.7 (17.11)
Baseline Area of Choroidal Neovascularization (CNV) [Mean (Standard Deviation); unit: mm^2] — SAF population used for analysis.
  mm^2 | 6.52 (5.245) [0 to 0] | 6.59 (5.052) [0 to 0] | 6.49 (4.437) [0 to 0] | 6.56 (5.129) [0 to 0] | 6.54 (4.968)
Baseline Lesion Type [Number; unit: patients] — SAF population used for analysis.
  patients
    Occult | 115 (0) [0 to 0] | 110 (0) [0 to 0] | 123 (0) [0 to 0] | 118 (0) [0 to 0] | 466
    Minimally Classic | 101 (0) [0 to 0] | 105 (0) [0 to 0] | 97 (0) [0 to 0] | 112 (0) [0 to 0] | 415
    Predominantly Classic | 82 (0) [0 to 0] | 87 (0) [0 to 0] | 82 (0) [0 to 0] | 71 (0) [0 to 0] | 322
    Missing | 6 (0) [0 to 0] | 2 (0) [0 to 0] | 2 (0) [0 to 0] | 2 (0) [0 to 0] | 12
Baseline Total Lesion Size [Mean (Standard Deviation); unit: mm^2] — SAF population used for analysis.
  mm^2 | 6.99 (5.491) [0 to 0] | 6.98 (5.388) [0 to 0] | 6.96 (4.711) [0 to 0] | 6.88 (5.214) [0 to 0] | 6.95 (5.202)
Baseline Best Corrected Visual Acuity (BCVA) [Mean (Standard Deviation); unit: letters read] — SAF population used for analysis. BCVA assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) chart. For BCVA tested via the 4 meter ETDRS protocol, 83 letters or more would represent 20/20 vision or better which would be considered an excellent outcome. Although, the ETDRS charts include 100 letters as the maximum possible score. The worst outcome is 0 letters read.
  letters read | 54.0 (13.43) [0 to 0] | 55.2 (13.15) [0 to 0] | 55.5 (13.12) [0 to 0] | 55.7 (12.84) [0 to 0] | 55.1 (13.14)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Maintained Vision at Week 52 - Last Observation Carried Forward (LOCF)
Description: Defined "maintenance of vision" as patients who lost fewer than 15 letters in Early Treatment Diabetic Retinopathy Study (ETDRS) letter score compared to baseline.
Time Frame: Baseline and at week 52
Population: PPS population used for analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Ranibizumab 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8 | Total
Number analyzed (Participants) | 269 | 285 | 270 | 265 | 1089
percentage of patients | 94.4 (0) | 95.1 (0) | 95.9 (0) | 95.1 (0) | 95.1 (0)
Statistical Analysis 1: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4; The statistical approach included a conditional sequence of calculations of the 95.1% CI using normal approximation of the difference between the proportion of patients with maintained vision at Week 52 for the group treated with 0.5 mg ranibizumab and the proportion of patients with maintained vision for each of the groups treated with IAI; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was set at 10%. The power is 90% according to the sample size estimation of the study protocol. Although not in the analysis plan for the study, in a separate communication, the FDA further explained that, whereas the 10% non-inferiority margin would be used to assess non-inferiority, a 5% non-inferiority margin would be used to assess clinical equivalence; Risk Difference (RD) = -0.7, 95.1% CI 2-sided [-4.4 to 3.1] — The difference is calculated as ranibizumab minus IAI. A positive value favors IAI 2.0Q4. As adjustment of multiple comparisons as conditional sequence of statistical hypotheses is used with alpha = 0.049
Statistical Analysis 2: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4; The statistical approach included a conditional sequence of calculations of the 95.1% CI using normal approximation of the difference between the proportion of patients with maintained vision at Week 52 for the group treated with 0.5 mg ranibizumab and the proportion of patients with maintained vision for each of the groups treated with IAI (EYLEA, VEGF Trap-Eye); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -1.5, 95.1% CI 2-sided [-5.1 to 2.1] — The difference is calculated as ranibizumab minus IAI. A negative value favors the IAI 0.5Q4 group. As adjustment of multiple comparisons as conditional sequence of statistical hypotheses is used with alpha = 0.049
Statistical Analysis 3: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.7, 95.1% CI 2-sided [-4.5 to 3.1] — The difference is calculated as ranibizumab minus IAI. A negative value favors the IAI 2.0Q8 group. As adjustment of multiple comparisons as conditional sequence of statistical hypotheses is used with alpha = 0.049

2. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) as Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score at Week 52 - LOCF
Description: Defined study baseline range of ETDRS Best Corrected Visual Acuity of: letter score of 73 to 25 (20/40 to 20/320) in the study eye; a higher score represents better functioning.
Time Frame: Baseline and at week 52
Population: FAS population used for analysis.
Measure: Mean (Standard Deviation); unit: letters read
Arm/Group | Ranibizumab 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8 | Total
Number analyzed (Participants) | 304 | 304 | 301 | 301 | 1210
letters read | 8.1 (15.25) | 10.9 (13.77) | 6.9 (13.41) | 7.9 (15.00) | 8.5 (14.44)
Statistical Analysis 1: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4; The pairwise comparison is performed as contrast statement in the analysis of covariance model with treatment group as fixed factor (all 4 treatment groups) and the baseline measure as covariate. The null hypothesis is that both mean changes are equal; Test type: Superiority or Other; p = 0.0054, ANCOVA — As adjustment of multiple comparisons, a conditional sequence of statistical hypotheses is used with alpha = 0.049; Differences in Least Squares means = 3.15, 95.1% CI 2-sided [0.92 to 5.37] — The difference is calculated as IAI minus ranibizumab. A positive value favors IAI 2.0Q4
Statistical Analysis 2: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4793, ANCOVA — As adjustment of multiple comparisons, a conditional sequence of statistical hypotheses is used with alpha = 0.049; Differences in Least Squares means = 0.80, 95.1% CI 2-sided [-3.03 to 1.43] — The difference is calculated as IAI minus ranibizumab. A positive value favors IAI 0.5Q4
Statistical Analysis 3: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8179, ANCOVA — As adjustment of multiple comparisons, a conditional sequence of statistical hypotheses is used with alpha = 0.049; Differences in Least Squares Means = 0.26, 95.1% CI 2-sided [-1.97 to 2.49] — The difference is calculated as IAI minus ranibizumab. A positive value favors IAI 2.0Q8

3. Secondary Outcome: Percentage of Patients Who Gained at Least 15 Letters of Vision in the ETDRS Letter Score in the Study Eye at Week 52 - LOCF.
Description: as for outcome 2
Time Frame: Baseline and at week 52
Population: FAS population used for analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Ranibizumab 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8 | Total
Number analyzed (Participants) | 304 | 304 | 301 | 301 | 1210
percentage of patients | 30.9 (0) | 37.5 (0) | 24.9 (0) | 30.6 (0) | 31.1 (0)
Statistical Analysis 1: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4; The null hypothesis is that both percentages are equal; Test type: Superiority or Other; p = 0.1042, Chi-squared — As adjustment of multiple comparisons, a conditional sequence of statistical hypotheses is used with alpha = 0.049; Risk Difference (RD) = 6.6, 95.1% CI 2-sided [-1.0 to 14.1] — The difference is calculated as IAI minus ranibizumab. A positive value favors IAI 2.0Q4
Statistical Analysis 2: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4; The null hypothesis is that both percentages are equal; Test type: Superiority or Other; p = 0.1037, Chi-squared — As adjustment of multiple comparisons, a conditional sequence of statistical hypotheses is used with alpha = 0.049; Risk Difference (RD) = -6.0, 95.1% CI 2-sided [-13.2 to 1.2] — The difference is calculated as IAI minus ranibizumab. A positive value favors IAI 0.5Q4
Statistical Analysis 3: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8; The pairwise The null hypothesis is that both percentages are equal; Test type: Superiority or Other; p = 0.93, Chi-squared — As adjustment of multiple comparisons, a conditional sequence of statistical hypotheses is used with alpha = 0.049; Risk Difference (RD) = -0.4, 95.1% CI 2-sided [-7.7 to 7.0] — The difference is calculated as VEGF Trap-Eye minus ranibizumab. A positive value favors VEGF Trap-Eye 2.0Q8

4. Secondary Outcome: Mean Change From Baseline in National Eye Institute Visual Functioning Questionnaire (NEI VFQ-25) Total Score at Week 52 - LOCF
Description: The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales which are all scored from 0-100. To reach the overall composite score, each sub-scale score is averaged in order to give each sub-scale equal weight.
Time Frame: Baseline and at Week 52
Population: FAS population used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ranibizumab 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8 | Total
Number analyzed (Participants) | 304 | 304 | 301 | 301 | 1210
scores on a scale | 4.9 (14.01) | 6.7 (13.50) | 4.5 (11.87) | 5.1 (14.74) | 5.3 (13.59)
Statistical Analysis 1: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2090, ANCOVA — As adjustment of multiple comparisons, a conditional sequence of statistical hypotheses is used with alpha = 0.049; Differences Least Squares means = 1.28, 95.1% CI 2-sided [-0.73 to 3.28] — The difference is calculated as IAI minus ranibizumab. A positive value favors IAI 2.0Q4
Statistical Analysis 2: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5128, ANCOVA — As adjustment of multiple comparisons, a conditional sequence of statistical hypotheses is used with alpha = 0.049; Differences in Least Squares means = -0.67, 95.1% CI 2-sided [-2.69 to 1.35] — The difference is calculated as IAI minus ranibizumab. A positive value favors IAI 0.5Q4
Statistical Analysis 3: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5579, ANCOVA — As adjustment of multiple comparisons, a conditional sequence of statistical hypotheses is used with alpha = 0.049; Differences in Least Squares means = -0.60, 95.1% CI 2-sided [-2.61 to 1.42] — The difference is calculated as IAI minus ranibizumab. A positive value favors IAI 2.0Q8

5. Secondary Outcome: Mean Change From Baseline in Choroidal Neovascularization (CNV) Area at Week 52 (LOCF)
Description: CNV area values measured in square millimeters (mm^2); lower values represent better outcomes.
Time Frame: Baseline and at week 52
Population: FAS population used for analysis.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Ranibizumab 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8 | Total
Number analyzed (Participants) | 304 | 304 | 301 | 301 | 1210
mm^2 | -4.2 (5.59) | -4.6 (5.47) | -3.5 (5.27) | -3.4 (6.02) | -3.9 (5.61)
Statistical Analysis 1: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3575, ANCOVA — As adjustment of multiple comparisons, a conditional sequence of statistical hypotheses is used with alpha = 0.049; Differences in Least Squares means = -0.33, 95.1% CI 2-sided [-1.04 to 0.38] — The difference is calculated as IAI minus ranibizumab. A negative value favors IAI 2.0Q4
Statistical Analysis 2: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0507, ANCOVA — As adjustment of multiple comparisons, a conditional sequence of statistical hypotheses is used with alpha = 0.049; Differences in Least Squares means = 0.71, 95.1% CI 2-sided [-0.01 to 1.42] — The difference is calculated as IAI minus ranibizumab. A negative value favors IAI 0.5Q4
Statistical Analysis 3: Comparison: Ranibizumab 0.5mg Q4 vs IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0173, ANCOVA — As adjustment of multiple comparisons, a conditional sequence of statistical hypotheses is used with alpha = 0.049; Differences in Least Squares means = 0.86, 95.1% CI 2-sided [0.15 to 1.58] — The difference is calculated as IAI minus ranibizumab. A negative value favors IAI 2.0Q8

ADVERSE EVENTS:
Time Frame: AEs reported from Day 1 to Wk 96. Yr 1 of tx (Day 1 to Wk 52): 21-day screening period followed by administration of study drug every 4 or 8 wks including sham injections at interim study visits (when study drug was not administered) for 48 wks.
Description: Yr 2 of tx (Wk 52 to Wk 96): Pts evaluated every 4 wks and received IVT injections of study drug (sham injections were not given) at intervals determined by specific re-treatment criteria. During this period, injections were given as frequently as every 4 weeks, but no less frequently than every 12 wks.
Groups:
- Ranibizumab 0.5mg Q4: Patients received a 0.5mg dose of ranibizumab via intravitreal (IVT) injection every 4 weeks for the first year. During the second year of treatment, patients were evaluated every 4 weeks and received IVT injections of ranibizumab (sham injections were not given) at intervals determined by specific re-treatment criteria. During this period, injections were given as frequently as every 4 weeks, but no less frequently than every 12 weeks.
- IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4: Patients received a 2.0mg dose of Intravitreal Aflibercept Injection (IAI, EYLEA, VEGF Trap-Eye) every 4 weeks for the first year. During the second year of treatment, patients were evaluated every 4 weeks and received IVT injections of Intravitreal Aflibercept Injection (IAI, EYLEA, VEGF Trap-Eye) (sham injections were not given) at intervals determined by specific re-treatment criteria. During this period, injections were given as frequently as every 4 weeks, but no less frequently than every 12 weeks.
- IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4: Patients received a 0.5mg dose of Intravitreal Aflibercept Injection (IAI, EYLEA, VEGF Trap-Eye) every 4 weeks for the first year. During the second year of treatment, patients were evaluated every 4 weeks and received IVT injections of Intravitreal Aflibercept Injection (IAI, EYLEA, VEGF Trap-Eye) (sham injections were not given) at intervals determined by specific re-treatment criteria. During this period, injections were given as frequently as every 4 weeks, but no less frequently than every 12 weeks.
- IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8: Patients received a 2.0mg dose of Intravitreal Aflibercept Injection (IAI, EYLEA, VEGF Trap-Eye) every 8 weeks (including one additional 2.0 mg dose at Week 4) for the first year and were to receive sham injections at interim monthly visits. During the second year of treatment, patients were evaluated every 4 weeks and received IVT injections of Intravitreal Aflibercept Injection (IAI, EYLEA, VEGF Trap-Eye) (sham injections were not given) at intervals determined by specific re-treatment criteria. During this period, injections were given as frequently as every 4 weeks, but no less frequently than every 12 weeks.
Arm/Group | Ranibizumab 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4 | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8
Serious Adverse Events (participants affected / at risk) | 94/304 | 70/304 | 88/304 | 90/303
Other Adverse Events (participants affected / at risk) | 261/304 | 254/304 | 262/304 | 258/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5mg Q4 (N=304) | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4 (N=304) | IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4 (N=304) | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8 (N=303)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 1 | 2
COAGULOPATHY (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
ATYPICAL FIBROXANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 1
BLADDER TRANSITIONAL CELL CARCINOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BREAST Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2
BREAST Neoplasms benign, malignant and unspecified (incl cysts and polyps) IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
BRONCHIOLOALVEOLAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
CARDIAC MYXOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
COLON Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
COLON Neoplasms benign, malignant and unspecified (incl cysts and polyps) RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
ENDOMETRIAL Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
HEPATIC Neoplasms benign, malignant and unspecified (incl cysts and polyps) METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2
LUNG SQUAMOUS CELL CARCINOMA STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
METASTASES TO Hepatobiliary disorders (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
NON-SMALL CELL LUNG Neoplasms benign, malignant and unspecified (incl cysts and polyps) METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
NON-SMALL CELL LUNG Neoplasms benign, malignant and unspecified (incl cysts and polyps) STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
PROSTATE Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 1
PROSTATE Neoplasms benign, malignant and unspecified (incl cysts and polyps) METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
RECTAL Neoplasms benign, malignant and unspecified (incl cysts and polyps) STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
RECTOSIGMOID Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
SALIVARY GLAND Neoplasms benign, malignant and unspecified (incl cysts and polyps) RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
SMALL CELL LUNG Neoplasms benign, malignant and unspecified (incl cysts and polyps) METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
SMALL CELL LUNG Neoplasms benign,malignant & unspecified(incl cysts and polyps)STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
SQUAMOUS CELL CARCINOMA OF Skin and subcutaneous tissue disorders (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3 | 2 | 4
THYROID Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
TONSIL Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
WALDENSTROM'S MACROGLOBULINAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
AORTIC ANEURYSM (Vascular disorders) | 1 | 2 | 1 | 0
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 1 | 0 | 0 | 0
AORTIC STENOSIS (Vascular disorders) | 1 | 1 | 2 | 1
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 1 | 1 | 2
FEMORAL ARTERY ANEURYSM (Vascular disorders) | 0 | 0 | 1 | 0
HAEMATOMA (Vascular disorders) | 0 | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 2 | 0 | 3 | 0
HYPOTENSION (Vascular disorders) | 0 | 1 | 0 | 0
ILIAC ARTERY OCCLUSION (Vascular disorders) | 0 | 0 | 1 | 0
LYMPHATIC FISTULA (Vascular disorders) | 1 | 0 | 0 | 0
LYMPHOCELE (Vascular disorders) | 1 | 0 | 0 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 0 | 0 | 1
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 0 | 1 | 0 | 0
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 1 | 0 | 0 | 1
PHLEBITIS (Vascular disorders) | 0 | 0 | 1 | 0
PHLEBITIS DEEP (Vascular disorders) | 0 | 1 | 0 | 0
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 | 0 | 0 | 1
MENIERE'S DISEASE (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 1 | 0 | 2
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0
ABDOMINAL HERNIA OBSTRUCTIVE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
COLITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 0 | 1 | 0
COLONIC POLYP (Gastrointestinal disorders) | 1 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0 | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0
FOOD POISONING (Gastrointestinal disorders) | 1 | 0 | 0 | 0
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 1
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 | 0 | 0 | 0
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 0 | 0 | 1 | 0
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ILEUS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 0 | 1 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 0 | 0 | 2 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 0 | 2 | 1
ASTHENIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
CATHETER SITE HAEMATOMA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
CHEST PAIN (Gastrointestinal disorders) | 2 | 1 | 2 | 0
DEATH (Gastrointestinal disorders) | 0 | 1 | 0 | 0
DEVICE DISLOCATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
DRUG WITHDRAWAL SYNDROME (Gastrointestinal disorders) | 0 | 0 | 1 | 0
NON-CARDIAC CHEST PAIN (Gastrointestinal disorders) | 1 | 1 | 0 | 0
PYREXIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
ACUTE CORONARY SYNDROME (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Ear and labyrinth disorders) | 1 | 2 | 2 | 1
ANGINA UNSTABLE (Ear and labyrinth disorders) | 3 | 0 | 0 | 0
AORTIC VALVE STENOSIS (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
ARRHYTHMIA (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
ARTERIOSCLEROSIS CORONARY ARTERY (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
ATRIAL FIBRILLATION (Ear and labyrinth disorders) | 3 | 2 | 7 | 7
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Ear and labyrinth disorders) | 0 | 0 | 0 | 0
BRADYCARDIA (Ear and labyrinth disorders) | 2 | 0 | 1 | 0
CARDIAC ARREST (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
CARDIAC FAILURE ACUTE (Ear and labyrinth disorders) | 1 | 0 | 2 | 0
CARDIAC FAILURE CHRONIC (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Ear and labyrinth disorders) | 4 | 2 | 4 | 8
CARDIO-RESPIRATORY ARREST (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
CARDIOMYOPATHY (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
CORONARY ARTERY DISEASE (Ear and labyrinth disorders) | 5 | 0 | 6 | 1
CORONARY ARTERY OCCLUSION (Ear and labyrinth disorders) | 1 | 2 | 0 | 0
CORONARY ARTERY STENOSIS (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
INTRACARDIAC THROMBUS (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
MITRAL VALVE INCOMPETENCE (Ear and labyrinth disorders) | 0 | 0 | 2 | 0
MYOCARDIAL INFARCTION (Ear and labyrinth disorders) | 6 | 1 | 5 | 2
MYOCARDIAL ISCHAEMIA (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
PERICARDIAL EFFUSION (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
SICK SINUS SYNDROME (Ear and labyrinth disorders) | 2 | 0 | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
TACHYARRHYTHMIA (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
TACHYCARDIA (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
VENTRICULAR FIBRILLATION (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
VENTRICULAR TACHYCARDIA (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0
ANORECTAL CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 0
ARTHRITIS BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 1
BACTERIAL DISEASE CARRIER (Infections and infestations) | 1 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 2 | 3
CELLULITIS (Infections and infestations) | 3 | 3 | 2 | 0
CLOSTRIDIAL Infections and infestationsION (Infections and infestations) | 0 | 1 | 0 | 2
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 0 | 1 | 0
DEVICE RELATED Infections and infestationsION (Infections and infestations) | 1 | 0 | 0 | 0
DIVERTICULITIS (Infections and infestations) | 1 | 1 | 0 | 1
ENCEPHALITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 1
ENDOCARDITIS (Infections and infestations) | 0 | 0 | 0 | 1
ESCHERICHIA URINARY TRACT Infections and infestationsION (Infections and infestations) | 1 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 1 | 0 | 2
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 1 | 1
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 1
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 1 | 0 | 0 | 0
LABYRINTHITIS (Infections and infestations) | 0 | 0 | 0 | 1
LOBAR PNEUMONIA (Infections and infestations) | 2 | 0 | 0 | 2
LUNG Infections and infestationsION (Infections and infestations) | 1 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 14 | 6 | 5 | 8
PYELONEPHRITIS (Infections and infestations) | 0 | 1 | 0 | 1
SCROTAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0
SEPSIS (Infections and infestations) | 0 | 0 | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 1 | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 0 | 1 | 0
SINUSITIS FUNGAL (Infections and infestations) | 0 | 0 | 1 | 0
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 0 | 1 | 1
UPPER RESPIRATORY TRACT Infections and infestationsION (Infections and infestations) | 0 | 0 | 0 | 0
URINARY TRACT Infections and infestationsION (Infections and infestations) | 1 | 3 | 0 | 0
URINARY TRACT Infections and infestationsION BACTERIAL (Infections and infestations) | 0 | 0 | 1 | 0
URINARY TRACT Infections and infestationsION STAPHYLOCOCCAL (Infections and infestations) | 0 | 0 | 1 | 0
UROSEPSIS (Infections and infestations) | 1 | 0 | 1 | 1
VESTIBULAR NEURONITIS (Infections and infestations) | 0 | 0 | 1 | 0
VIRAL Infections and infestationsION (Infections and infestations) | 0 | 0 | 1 | 0
VIRAL PERICARDITIS (Infections and infestations) | 1 | 0 | 0 | 0
WOUND Infections and infestationsION BACTERIAL (Infections and infestations) | 0 | 1 | 0 | 0
ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 8 | 13 | 7 | 16
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
HEAD Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 4 | 2 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 0
INCISIONAL HERNIA, OBSTRUCTIVE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
JOINT Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
MENISCUS LESION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
POST LAMINECTOMY SYNDROME (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
SNAKE BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 2
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
TRAUMATIC BRAIN Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood and lymphatic system disorders GLUCOSE INCREASED (Investigations) | 0 | 1 | 0 | 0
Blood and lymphatic system disorders PRESSURE INCREASED (Investigations) | 0 | 0 | 0 | 1
Blood and lymphatic system disorders PRESSURE ORTHOSTATIC ABNORMAL (Investigations) | 0 | 0 | 1 | 0
CALCULUS BLADDER (Renal and urinary disorders) | 0 | 0 | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 0 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 0 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 3 | 2 | 2
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 1 | 0 | 0 | 0
BILE DUCT STONE (Hepatobiliary disorders) | 1 | 0 | 0 | 1
CHOLANGITIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 2
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 0 | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 | 1 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 1 | 2 | 0
PORTAL HYPERTENSION (Hepatobiliary disorders) | 0 | 0 | 1 | 0
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
SHOCK HYPOGLYCAEMIC (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
APHASIA (Nervous system disorders) | 0 | 1 | 0 | 0
BALANCE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 1
CAROTID ARTERY DISEASE (Nervous system disorders) | 0 | 0 | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 2 | 0 | 0
CEREBELLAR INFARCTION (Nervous system disorders) | 1 | 0 | 0 | 0
CEREBRAL ARTERY THROMBOSIS (Nervous system disorders) | 0 | 1 | 0 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 1 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 0 | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 | 3 | 1 | 5
COMA (Nervous system disorders) | 1 | 0 | 0 | 0
CONVULSION (Nervous system disorders) | 0 | 0 | 0 | 1
DEMENTIA (Nervous system disorders) | 0 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 1 | 0 | 1
EMBOLIC STROKE (Nervous system disorders) | 1 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1 | 0 | 0
LACUNAR INFARCTION (Nervous system disorders) | 1 | 1 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 0 | 0
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 0 | 1 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 1 | 1 | 1
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 0 | 1 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 1 | 1
SYNCOPE (Nervous system disorders) | 3 | 1 | 3 | 1
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 0 | 0 | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 3 | 7 | 5
CHOLECYSTECTOMY (Surgical and medical procedures) | 0 | 1 | 0 | 0
MICROGRAPHIC Skin and subcutaneous tissue disorders SURGERY (Surgical and medical procedures) | 0 | 0 | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 2 | 0 | 0 | 1
Psychiatric disordersOTIC DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 1
CYSTOCELE (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
RECTOCELE (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
APNOEIC ATTACK (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 6 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
RESTRICTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
TRACHEAL MASS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
AGE-RELATED MACULAR DEGENERATION (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Fellow Eye disorders
BLEPHARITIS (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Fellow Eye disorders
CATARACT (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Fellow Eye disorders
CHOROIDAL NEOVASCULARISATION (Eye disorders) | 1 | 0 | 0 | 0 — Ocular Fellow Eye disorders
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Fellow Eye disorders
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 0 | 1 — Ocular Fellow Eye disorders
MACULAR DEGENERATION (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Fellow Eye disorders
MACULOPATHY (Eye disorders) | 0 | 0 | 1 | 0 — Ocular Fellow Eye disorders
POSTERIOR CAPSULE OPACIFICATION (Eye disorders) | 1 | 0 | 0 | 0 — Ocular Fellow Eye disorders
RETINAL DETACHMENT (Eye disorders) | 0 | 0 | 2 | 0 — Ocular Fellow Eye disorders
RETINAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 1 — Ocular Fellow Eye disorders
RETINAL OEDEMA (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Fellow Eye disorders
RETINAL TEar and labyrinth disorders (Eye disorders) | 0 | 0 | 0 | 1 — Ocular Fellow Eye disorders
UVEITIS (Eye disorders) | 0 | 0 | 0 | 1 — Ocular Fellow Eye disorders
VISUAL ACUITY REDUCED (Eye disorders) | 1 | 1 | 3 | 0 — Ocular Fellow Eye disorders
VITREOUS DETACHMENT (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Fellow Eye disorders
ENDOPHTHALMITIS (Infections and infestations) | 1 | 0 | 1 | 0 — Ocular Fellow Eye disorders
INTRAOCULAR PRESSURE INCREASED (Investigations) | 0 | 0 | 0 | 0 — Ocular Fellow Eye disorders
ANGLE CLOSURE GLAUCOMA (Eye disorders) | 0 | 1 | 0 | 0 — Ocular Study Eye disorders
BLINDNESS TRANSIENT (Eye disorders) | 1 | 0 | 0 | 0 — Ocular Study Eye disorders
CHOROIDAL HAEMORRHAGE (Eye disorders) | 1 | 0 | 0 | 0 — Ocular Study Eye disorders
DRY Eye disorders (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Study Eye disorders
Eye disorders IRRITATION (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Study Eye disorders
Eye disorders PAIN (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Study Eye disorders
Eye disorders PRURITUS (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Study Eye disorders
FOREIGN BODY SENSATION IN Eye disordersS (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Study Eye disorders
KERATITIS (Eye disorders) | 0 | 1 | 0 | 0 — Ocular Study Eye disorders
LACRIMATION INCREASED (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Study Eye disorders
MACULAR HOLE (Eye disorders) | 0 | 0 | 1 | 0 — Ocular Study Eye disorders
PSEUDOENDOPHTHALMITIS (Eye disorders) | 1 | 0 | 0 | 0 — Ocular Study Eye disorders
RETINAL DEGENERATION (Eye disorders) | 0 | 1 | 0 | 0 — Ocular Study Eye disorders
RETINAL PIGMENT EPITHELIAL TEar and labyrinth disorders (Eye disorders) | 0 | 0 | 0 | 1 — Ocular Study Eye disorders
RETINAL PIGMENT EPITHELIOPATHY (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Study Eye disorders
VISION BLURRED (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Study Eye disorders
VITREOUS FLOATERS (Eye disorders) | 0 | 0 | 0 | 0 — Ocular Study Eye disorders
VITREOUS HAEMORRHAGE (Eye disorders) | 1 | 0 | 0 | 0 — Ocular Study Eye disorders
INCORRECT DOSE ADMINISTERED (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — Ocular Study Eye disorders
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5mg Q4 (N=304) | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q4 (N=304) | IAI (EYLEA, VEGF Trap-Eye) 0.5mg Q4 (N=304) | IAI (EYLEA, VEGF Trap-Eye) 2.0mg Q8 (N=303)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 17 | 18 | 17 | 8
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 | 14 | 13 | 16
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 11 | 15 | 17
HYPERTENSION (Vascular disorders) | 35 | 30 | 32 | 33
DIARRHOEA (Gastrointestinal disorders) | 18 | 18 | 8 | 9
NAUSEA (Gastrointestinal disorders) | 15 | 16 | 15 | 15
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Ear and labyrinth disorders) | 16 | 18 | 8 | 9
BRONCHITIS (Infections and infestations) | 23 | 19 | 16 | 24
NASOPHARYNGITIS (Infections and infestations) | 36 | 46 | 41 | 39
SINUSITIS (Infections and infestations) | 18 | 13 | 17 | 14
UPPER RESPIRATORY TRACT Infections and infestationsION (Infections and infestations) | 18 | 18 | 19 | 26
URINARY TRACT Infections and infestationsION (Infections and infestations) | 26 | 22 | 25 | 23
FALL (Injury, poisoning and procedural complications) | 19 | 13 | 15 | 21
Blood and lymphatic system disorders GLUCOSE INCREASED (Investigations) | 13 | 12 | 17 | 16
HEADACHE (Nervous system disorders) | 21 | 14 | 16 | 15
COUGH (Respiratory, thoracic and mediastinal disorders) | 16 | 13 | 10 | 13
AGE-RELATED MACULAR DEGENERATION (Eye disorders) | 21 | 16 | 12 | 15 — Ocular Fellow Eye disorders
BLEPHARITIS (Eye disorders) | 16 | 18 | 14 | 14 — Ocular Fellow Eye disorders
CATARACT (Eye disorders) | 10 | 17 | 10 | 10 — Ocular Fellow Eye disorders
CHOROIDAL NEOVASCULARISATION (Eye disorders) | 17 | 10 | 13 | 9 — Ocular Fellow Eye disorders
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 16 | 17 | 16 | 19 — Ocular Fellow Eye disorders
MACULAR DEGENERATION (Eye disorders) | 22 | 14 | 21 | 14 — Ocular Fellow Eye disorders
RETINAL HAEMORRHAGE (Eye disorders) | 43 | 36 | 36 | 22 — Ocular Fellow Eye disorders
RETINAL OEDEMA (Eye disorders) | 18 | 8 | 12 | 11 — Ocular Fellow Eye disorders
VISUAL ACUITY REDUCED (Eye disorders) | 27 | 10 | 20 | 19 — Ocular Fellow Eye disorders
VITREOUS DETACHMENT (Eye disorders) | 16 | 24 | 25 | 24 — Ocular Fellow Eye disorders
INTRAOCULAR PRESSURE INCREASED (Investigations) | 16 | 8 | 15 | 15 — Ocular Fellow Eye disorders
DRY Eye disorders (Eye disorders) | 12 | 16 | 10 | 14 — Ocular Study Eye disorders
Eye disorders IRRITATION (Eye disorders) | 19 | 13 | 15 | 16 — Ocular Study Eye disorders
Eye disorders PAIN (Eye disorders) | 34 | 39 | 35 | 31 — Ocular Study Eye disorders
Eye disorders PRURITUS (Eye disorders) | 11 | 16 | 10 | 6 — Ocular Study Eye disorders
FOREIGN BODY SENSATION IN Eye disordersS (Eye disorders) | 9 | 10 | 10 | 19 — Ocular Study Eye disorders
LACRIMATION INCREASED (Eye disorders) | 11 | 11 | 15 | 16 — Ocular Study Eye disorders
RETINAL PIGMENT EPITHELIOPATHY (Eye disorders) | 14 | 18 | 17 | 14 — Ocular Study Eye disorders
VISION BLURRED (Eye disorders) | 12 | 18 | 17 | 13 — Ocular Study Eye disorders
VITREOUS FLOATERS (Eye disorders) | 47 | 49 | 30 | 29 — Ocular Study Eye disorders

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After completion of the trial, the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review; provided that the sponsor can remove confidential or proprietary information from such communications. The sponsor cannot require other changes to the communication and cannot extend the embargo.